## The Safety, Efficacy and Pharmacokinetics of Dexmedetomidine Administered Through Different Routes in Pediatric

**October 12, 2017** 

## **Statistical Analysis Plan**

All data are presented as mean  $\pm$  SD, median (interquartile range) or number (%), as appropriate. The normal distribution of data was examined with one-factor ANOVA and Fisher's-LSD test. Fisher exact Chi-square test was used to compare gender, surgery types, weight, bradycardia,ED and supplementary drugs in PACU and so on. HR,MBP,and duration of surgery and so on were examined with Mann-Whitney U test. Data were analyzed using SPSS software (SPSS 16.0, SPSS, Inc., Chicago, IL, USA). A p value less than 0.05 was considered as to be a significant difference.